CLINICAL TRIAL: NCT05191342
Title: The Expression of Proprotein Convertase Subtilisin Kexin 9 in Patients With Rheumatoid Arthritis Combined Atrial Fibrillation
Brief Title: Proprotein Convertase Subtilisin Kexin 9 in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Other Study IDs: Atrial fibrillation and RA
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: PCSK9
Keywords: Atrial fibrillation; Rheumatoid arthritis; PCSK9
MeSH Terms: conditions — Atrial Fibrillation; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: Patients with rheumatoid arthritis (n=25).
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay for PCSK9
- Rheumatoid arthritis complicated atrial fibrillation: Patients with rheumatoid arthritis complicated atrial fibrillation (n=25).
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay for PCSK9
- healthy volunteers: Healthy volunteers (n=25).
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay for PCSK9

INTERVENTIONS:
Diagnostic Test: Enzyme-linked immunosorbent assay for PCSK9 — Enzyme-linked immunosorbent assay for plasma PCSK9

SUMMARY:
Rheumatoid arthritis (RA) has been proved to increase the incidence of atrial fibrillation (AF) with persistent systemic inflammation. Proprotein convertase subtilisin/kexin type 9 (PCSK9) has been found to enhance the production of pro-inflammatory cytokines. Therefore, we performed the present study to observe the expression and significance of proprotein convertase subtilisin kexin 9 (PCSK9) in patients with RA combined atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), the most common clinically relevant arrhythmia, is an important contributor to population morbidity and mortality. Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease, which affects approximately 1% of the population. Increasing studies demonstrated that RA had a positive correlation with increased cardiovascular diseases. Increasing studies showed that the prevalence of AF is significantly higher in RA patients than in the general population. Recently, some studies indicated that proprotein convertase subtilisin/kexin type 9 (PCSK9) promotes inflammatory by regulating macrophage secretion of inflammatory cytokines, inducing C-reaction protein (CRP), interleukin (IL)-6, IL-8, tumor necrosis factor-α (TNF-α) and so on. However, the levels of PCSK9 in atrial fibrillation patients with rheumatoid arthritis is still unclear. Therefore, the aim of this study was to assess the expression of PCSK9 in patients with RA combined atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Rheumatoid arthritis
2. Rheumatoid arthritis combined with AF

Exclusion Criteria:

1. (1) History of hypertension, diabetes, cardiovascular disease, severe impairment of liver function, severe renal insufficiency.

(2) Infectious diseases. (3) History malignant tumor. (4) Pregnant women, Lactating women. (5) Other autoimmune diseases.

2. (1) History of hypertension, diabetes, cardiovascular disease (except for AF), severe impairment of liver function, severe renal insufficiency.

(2) Infectious diseases. (3) History malignant tumor. (4) Pregnant women, Lactating women. (5) Other autoimmune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis (n=25), patients with rheumatoid arthritis complicated atrial fibrillation (n=25) and healthy volunteers (n=25). ELISA were used to test plasma PCSK9.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The expression of PCSK9 in patients with RA combined with AF | One year
  To assess the expression and significance of plasma PCSK9 in three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, Doctor, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (2):
- China (2):
  - the first affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Thrombelastogram, Harbin, Heilongjiang